CLINICAL TRIAL: NCT01047345
Title: A Phase III, Randomized, International, Placebo-Controlled, Double-Blind Clinical Trial to Study the Tolerability and Immunogenicity of V503, a Multivalent Human Papillomavirus (HPV) L1 Virus-Like Particle (VLP) Vaccine, Given to Females 12-26 Years of Age Who Have Previously Received GARDASIL™
Brief Title: A Study of V503, a 9-valent Human Papillomavirus (9vHPV) Vaccine in Females 12-26 Years of Age Who Have Previously Received GARDASIL™ (V503-006)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V503-006; 2010_504 (Other: Merck Registration Number)
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Results first posted 2014-12-22 (Estimated); Last update posted 2018-11-27 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancers; Vulvar Cancers; Vaginal Cancers; Genital Warts
Keywords: Cervical cancer; Genital warts; Human papillomavirus vaccine; GARDASIL™
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 9vHPV Vaccine (Experimental): Blinded 9vHPV vaccine (V503) 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6 of the Base Study. Participants will not continue to the Extension Study.
  Interventions: Biological: V503
- Placebo (Placebo Comparator): Blinded 0.5 mL intramuscular injection of saline placebo at Day 1, Month 2, and Month 6 of the Base Study. After completion of the Base Study, participants will be eligible to receive open-label 9vHPV 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6 of the Extension Study.
  Interventions: Biological: V503; Biological: Placebo to V503

INTERVENTIONS:
Biological: V503 — V503 (9vHPV) vaccine given as a 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6 of the Base Study or the Study Extension
Biological: Placebo to V503 — Placebo to V503 (saline) given as a 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6 of the Base Study
  Arms: Placebo

SUMMARY:
This study will evaluate whether V503 (9vHPV vaccine), is well tolerated in girls and women between 12 and 26 years old who have previously been vaccinated with GARDASIL™. Participants will receive vaccination with 9vHPV vaccine or placebo on Day 1, Month 2, and Month 6 of the Base Study. Participants who receive placebo in the Base Study will be eligible to receive vaccination with 9vHPV vaccine on Day 1, Month 2, and Month 6 of the Extension Study.

ELIGIBILITY:
Inclusion Criteria:

Participants Age 12 to 15 Years:

* Participant is in good health
* Parent/legal guardian and participant agree to provide study personnel with a primary telephone number for follow-up
* Participant received a 3-dose regimen of marketed GARDASIL™ within a 1 year period and the last dose of GARDASIL™ was at least 1 year from study day 1
* Participant has not received any other HPV vaccine
* Participant is not yet sexually active

Participants Age 16 to 26 Years:

* Participant is in good health
* Participant agrees to provide a primary telephone number for follow-up
* Participant received a 3-dose regimen of marketed GARDASIL™ within a 1 year period and the last dose of GARDASIL™ was at least 1 year from study day 1
* Participant has not received any other HPV vaccine
* Participant has never had Papanicolaou (Pap) testing or has only had normal results
* Participant has a history of 0 to 4 lifetime sexual partners at enrollment

Exclusion Criteria:

All participants:

* Participant has a history of severe allergic reaction that required medical intervention
* Participant has any disorder that would contraindicate intramuscular injections
* Participant is pregnant
* Participant is immunocompromised or has an autoimmune condition
* Participant has had a splenectomy
* Participant has received any immune globulin product or blood-derived product
* Participant has participated in a HPV vaccine clinical trial

Participants Age 16 to 26 Only:

* Participant expects to donate eggs during the study
* Participant has a history of abnormal cervical biopsy result
* Participant has a history of HPV-related external genital lesions, external genital cancer, HPV-related vaginal lesions, or vaginal cancer

Ages: 12 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 924 (Actual)
Dates: Start 2010-02-24 (Actual); Primary Completion 2011-06-10 (Actual); Study Completion 2015-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Garland SM, Cheung TH, McNeill S, Petersen LK, Romaguera J, Vazquez-Narvaez J, Bautista O, Shields C, Vuocolo S, Luxembourg A. Safety and immunogenicity of a 9-valent HPV vaccine in females 12-26 years of age who previously received the quadrivalent HPV vaccine. Vaccine. 2015 Nov 27;33(48):6855-64. doi: 10.1016/j.vaccine.2015.08.059. Epub 2015 Sep 26. PMID 26411885
- [Result] Moreira ED Jr, Block SL, Ferris D, Giuliano AR, Iversen OE, Joura EA, Kosalaraksa P, Schilling A, Van Damme P, Bornstein J, Bosch FX, Pils S, Cuzick J, Garland SM, Huh W, Kjaer SK, Qi H, Hyatt D, Martin J, Moeller E, Ritter M, Baudin M, Luxembourg A. Safety Profile of the 9-Valent HPV Vaccine: A Combined Analysis of 7 Phase III Clinical Trials. Pediatrics. 2016 Aug;138(2):e20154387. doi: 10.1542/peds.2015-4387. Epub 2016 Jul 15. PMID 27422279
- [Derived] Moreira ED, Giuliano AR, de Hoon J, Iversen OE, Joura EA, Restrepo J, Van Damme P, Vandermeulen C, Ellison MC, Krick A, Shields C, Heiles B, Luxembourg A. Safety profile of the 9-valent human papillomavirus vaccine: assessment in prior quadrivalent HPV vaccine recipients and in men 16 to 26 years of age. Hum Vaccin Immunother. 2018 Feb 1;14(2):396-403. doi: 10.1080/21645515.2017.1403700. Epub 2017 Dec 14. PMID 29211620
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V503-006&kw=V503-006&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- 9vHPV Vaccine - Base Study: Blinded 9vHPV vaccine (V503) 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6 of the Base Study. Participants will not continue to the Extension Study.
- Placebo - Base Study: Blinded 0.5 mL intramuscular injection of saline placebo at Day 1, Month 2, and Month 6 of the Base Study. After completion of the Base Study, participants will be eligible to receive open-label 9vHPV 0.5 mL intramuscular injection at Day 1, Month 2, and Month 6 of the Extension Study.
- 9vHPV Vaccine - Extension Study: Participants who received placebo in Base Study and elected to have open-label 9vHPV vaccination in Extension Study.
Period: Base Study
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study | 9vHPV Vaccine - Extension Study
Started | 618 | 306 | 0
Vaccination 1 | 615 | 306 | 0
Vaccination 2 | 604 | 304 | 0
Vaccination 3 | 597 | 300 | 0
Completed | 596 (Includes 1 participant for whom completion status is unknown) | 300 | 0
Not Completed | 22 | 6 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Lost to Follow-up | 4 | 1 | 0
Not completed — Protocol Violation | 3 | 1 | 0
Not completed — Withdrawal by Subject | 12 | 4 | 0
Period: Extension
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study | 9vHPV Vaccine - Extension Study
Started | 0 | 0 | 102 (Not all eligible participants elected to participate in extension)
Vaccination 4 | 0 | 0 | 102
Vaccination 5 | 0 | 0 | 99
Vaccination 6 | 0 | 0 | 95 (1 participant received 6th vaccination outside the context of study but completed the study.)
Completed | 0 | 0 | 96
Not Completed | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study | Total
Number analyzed (Participants) | 618 | 306 | 924
Age, Customized [Number; unit: Participants]
  12 to 15 years | 122 | 60 | 182
  16 to 26 years | 496 | 246 | 742
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 618 | 306 | 924
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience an Injection-site Adverse Event (AE) - Base Study
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. The percentage of participants who reported an AE that was associated with the injection site such as redness, swelling, and pain/tenderness/soreness was summarized.
Time Frame: up to 5 days after any vaccination - Base Study
Population: All participants who received at least 1 vaccination and had available follow-up data.
Measure: Number; unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study
Number analyzed (Participants) | 608 | 305
Percentage of Participants | 91.1 | 43.9

2. Primary Outcome: Percentage of Participants With Body Temperature ≥100.0°F (≥37.8ºC) - Base Study
Description: Participants collected their oral body temperature in the evening of their vaccination day and at the same time each day thereafter for 4 days. The maximum body temperature obtained within 5 days of any of the 3 vaccinations was recorded.
Time Frame: up to 5 days after any vaccination - Base Study
Population: All participants who received at least 1 vaccination and had available temperature data.
Measure: Number; unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study
Number analyzed (Participants) | 604 | 304
Percentage of Participants | 6.5 | 3.0
Statistical Analysis 1: Comparison: 9vHPV Vaccine - Base Study vs Placebo - Base Study; Test type: Superiority or Other; p = 0.026, Miettinen & Nurminen; Difference in Percentages = 3.5, 95% CI 2-sided [0.5 to 6.2]

3. Primary Outcome: Percentage of Participants Who Experience a Systemic AE - Base Study
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Systemic AEs were those not categorized as injection-site AEs.
Time Frame: up to 14 days after any vaccination - Base Study
Population: All participants who received at least 1 vaccination and had available follow-up data.
Measure: Number; unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study
Number analyzed (Participants) | 608 | 305
Percentage of Participants | 59.7 | 55.7
Statistical Analysis 1: Comparison: 9vHPV Vaccine - Base Study vs Placebo - Base Study; Test type: Superiority or Other; Miettinen & Nurminen; Difference in Percentages = 4.0, 95% CI 2-sided [-2.8 to 10.8]

4. Primary Outcome: Percentage of Participants Who Experience a Serious Adverse Event (SAE) Within 15 Days of Any Vaccination - Base Study
Description: An SAE is one that results in death, disability/incapacity, or hospitalization or is life threatening, a congenital anomaly or birth defect, cancer, an overdose, or otherwise jeopardizes the participant and may require medical intervention.
Time Frame: up to 14 days after any vaccination - Base Study
Population: All participants who received at least 1 vaccination and had available follow-up data.
Measure: Number; unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study
Number analyzed (Participants) | 608 | 305
Percentage of Participants | 0.3 | 0.3
Statistical Analysis 1: Comparison: 9vHPV Vaccine - Base Study vs Placebo - Base Study; Test type: Superiority or Other; Miettinen & Nurminen; Difference in Percentages = 0.0, 95% CI 2-sided [-1.5 to 0.9]

5. Primary Outcome: Percentage of Participants Who Experience a Vaccine-related SAE Any Time During Study- Base Study
Description: An SAE is one that results in death, disability/incapacity, or hospitalization or is life threatening, a congenital anomaly or birth defect, cancer, an overdose, or otherwise jeopardizes the participant and may require medical intervention. An SAE that is judged by the Investigator to be "definitely related," "probably related," or "possibly related" is defined as a vaccine-related SAE.
Time Frame: Up to 7 months - Base Study
Population: All participants who received at least 1 vaccination and had available follow-up data.
Measure: Number; unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study
Number analyzed (Participants) | 608 | 305
Percentage of Participants | 0.2 | 0.3
Statistical Analysis 1: Comparison: 9vHPV Vaccine - Base Study vs Placebo - Base Study; Test type: Superiority or Other; Miettinen & Nurminen; Difference in Percentages = -0.2, 95% CI 2-sided [-1.7 to 0.6]

6. Primary Outcome: Percentage of Participants Who Experience a Severe Injection-site AE - Base Study
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Participants were instructed to estimate the severity of AEs such as pain at injection site as mild (awareness of symptom, but easily tolerated), moderate (discomfort enough to cause interference with usual activities), or severe (incapacitating with inability to work or do usual activity). Additionally, participants were instructed to measure any swelling and/or erythema at its greatest width. Swelling or erythema with diameter >2 inches (>5 cm) was recorded as severe. All AEs associated with the injection site and reported as severe were summarized.
Time Frame: up to 5 days after any vaccination - Base Study
Population: All participants who received at least 1 vaccination and had available follow-up data.
Measure: Number; unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study
Number analyzed (Participants) | 608 | 305
Percentage of Participants | 11.2 | 1.0
Statistical Analysis 1: Comparison: 9vHPV Vaccine - Base Study vs Placebo - Base Study; Test type: Superiority or Other; Miettinen & Nurminen; Difference in Percentages = 10.2, 95% CI 2-sided [7.5 to 13.1]

7. Secondary Outcome: Percentage of Participants Who Seroconvert to Each of the HPV Types Contained in the Vaccine - Base Study
Description: Serum antibody titers for HPV virus-like particles (VLPs), Types 6, 11, 16, 18, 31, 33, 45, 52 and 58 were determined 4 weeks post-vaccination 3 using competitive luminex immunoassay (cLIA). The serostatus cutoffs (milli Merck U/mL) for HPV types were as follows: HPV Type 6: ≥30, HPV Type 11: ≥16; HPV Type 16: ≥20, HPV Type 18: ≥24, HPV Type 31: ≥10, HPV Type 33: ≥8, HPV Type 45: ≥8, HPV Type 52: ≥8, and HPV Type 58: ≥8.
Time Frame: 4 weeks post-vaccination 3 (Month 7; End of Base Study)
Population: Participants who received all 3 vaccinations within an acceptable day range, had Month 7 serology sample collected within an acceptable range and had no other protocol violations that could interfere with immunes response to the vaccine. Statistical testing performed only within the 9vHPV arm and only for HPV types 31, 33, 45, 52, and 58.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study
Number analyzed (Participants) | 515 | 261
Percentage of Participants
  Anti-HPV 6 (n=511; n=251) | 100.0 [99.3 to 100.0] | 100.0 [98.5 to 100.0]
  Anti-HPV 11 (n=515; n=261) | 100.0 [99.3 to 100.0] | 99.6 [97.9 to 100.0]
  Anti-HPV 16 (n=515; n=261) | 100.0 [99.3 to 100.0] | 100.0 [98.6 to 100.0]
  Anti-HPV 18 (n=515; n=261) | 100.0 [99.3 to 100.0] | 85.4 [80.6 to 89.5]
  Anti-HPV 31 (n=515; n=261) | 99.8 [98.9 to 100.0] | 23.8 [18.7 to 29.4]
  Anti-HPV 33 (n=515; n=261) | 99.8 [98.9 to 100.0] | 8.0 [5.0 to 12.0]
  Anti-HPV 45 (n=515; n=261) | 98.3 [96.7 to 99.2] | 3.4 [1.6 to 6.4]
  Anti-HPV 52 (n=515; n=261) | 99.6 [98.6 to 100.0] | 3.8 [1.9 to 6.9]
  Anti-HPV 58 (n=515; n=261) | 99.8 [98.9 to 100.0] | 9.2 [6.0 to 13.4]
Statistical Analysis 1: Comparison: 9vHPV Vaccine - Base Study; Anti-HPV 31; Test type: Superiority or Other; p < 0.001, Clopper-Pearson — statistical criterion of acceptability required that the lower bound of the 95% confidence interval (CI) for the proportion of participants seroconverting be greater than 90%; Seroconversion rate = 99.8, 95% CI 2-sided [98.9 to 100.0]
Statistical Analysis 2: Comparison: 9vHPV Vaccine - Base Study; Anti-HPV 33; Test type: Superiority or Other; p < 0.001, Clopper-Pearson — statistical criterion of acceptability required that the lower bound of the 95% CI for the proportion of subjects seroconverting be greater than 90%; Seroconversion Rate = 99.8, 95% CI 2-sided [98.9 to 100.0]
Statistical Analysis 3: Comparison: 9vHPV Vaccine - Base Study; Anti-HPV 45; Test type: Superiority or Other; p < 0.001, Clopper-Pearson — [p-value comment as in outcome 7, analysis 2]; Seroconversion Rate = 98.3, 95% CI 2-sided [96.7 to 99.2]
Statistical Analysis 4: Comparison: 9vHPV Vaccine - Base Study; Anti-HPV 52; Test type: Superiority or Other; p < 0.001, Clopper-Pearson — [p-value comment as in outcome 7, analysis 2]; Seroconversion Rate = 99.6, 95% CI 2-sided [98.6 to 100.0]
Statistical Analysis 5: Comparison: 9vHPV Vaccine - Base Study; Anti-HPV 58; Test type: Superiority or Other; p < 0.001, Clopper-Pearson — [p-value comment as in outcome 7, analysis 2]; Seroconversion Rate = 99.8, 95% CI 2-sided [98.9 to 100.0]

8. Other Pre Specified Outcome: Percentage of Participants Who Experience an SAE- Extension Study
Description: as for outcome 4
Time Frame: up to Month 7 - Extension Study
Population: All participants who received at least 1 vaccination in Extension Study and had available follow-up data.
Measure: Number; unit: Percentage of Participants
Arm/Group | 9vHPV Vaccine - Extension Study
Number analyzed (Participants) | 99
Percentage of Participants | 2.0

ADVERSE EVENTS:
Time Frame: Up to 5 days after any vaccination (Non-serious injection site AEs); up to 15 days after any vaccination (Non-serious systemic AEs) and up to 7 months (Serious AEs) - Base Study and Extension Study
Description: Population included all participants who received at least 1 vaccination and had available follow-up data. Only SAEs were collected systematically in the Extension Study. Although some unsolicited non-serious AEs were reported during the Extension Study, none exceeded the 5% cut-off.
Arm/Group | 9vHPV Vaccine - Base Study | Placebo - Base Study | 9vHPV Vaccine - Extension Study
Serious Adverse Events (participants affected / at risk) | 3/608 | 3/305 | 2/99
Other Adverse Events (participants affected / at risk) | 566/608 | 197/305 | 0/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9vHPV Vaccine - Base Study (N=608) | Placebo - Base Study (N=305) | 9vHPV Vaccine - Extension Study (N=99)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 9vHPV Vaccine - Base Study (N=608) | Placebo - Base Study (N=305) | 9vHPV Vaccine - Extension Study (N=99)
Nausea (Gastrointestinal disorders) | 52 (67) | 12 (13) | 0 (0)
Injection site erythema (General disorders) | 258 (420) | 26 (33) | 0 (0)
Injection site pain (General disorders) | 549 (1392) | 117 (182) | 0 (0)
Injection site pruritus (General disorders) | 48 (68) | 4 (5) | 0 (0)
Injection site swelling (General disorders) | 298 (558) | 18 (27) | 0 (0)
Pyrexia (General disorders) | 42 (50) | 10 (10) | 0 (0)
Nasopharyngitis (Infections and infestations) | 47 (55) | 19 (20) | 0 (0)
Dizziness (Nervous system disorders) | 31 (34) | 6 (8) | 0 (0)
Headache (Nervous system disorders) | 190 (318) | 81 (150) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 40 (46) | 12 (14) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.